CLINICAL TRIAL: NCT05357625
Title: The Impact of Feedback Informed Treatment in Floating Support Service - a Randomized Controlled Trial
Brief Title: The Impact of Feedback Informed Treatment in Floating Support Service
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: Copenhagen Municipality, Denmark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SFI 2808
Record Dates: First submitted 2016-07-08; First posted 2022-05-03 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2016-07

CONDITIONS: Quality of Life
Keywords: Partners for change outcome management system; Feedback-informed treatment; Routine Outcome management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Clients in the treatment group received the usual floating support service as described for the control group together with feedback. The support workers received feedback from the clients through the ORS and SRS scales of the feedback tool (Bargmann and Robinson 2011). The support worker evaluated the progress of the outcome for the client and the alliance between the support worker and the client from session to session.
  Interventions: Behavioral: Feedback Informed Treatment
- Control group (No Intervention): Clients in the control group received the usual floating support service without Feedback. Therefore, there was no systematic feedback between clients and support workers in the control group. The service was provided in the clients' homes, and there was no fixed limit of sessions for the support. The support covered any problem, including setting up tenancies, working with clients around practical things, so they could live independently, making sure that clients received all relevant benefits and helping clients with access to physical and mental health services. Some support workers saw their clients on a weekly basis, but there was a large variation in the frequency of meetings. Furthermore, the duration of the support service varied, from a few weeks to several years.

INTERVENTIONS:
Behavioral: Feedback Informed Treatment — FIT is based on two simple questionnaires and aims to assess and improve the effectiveness of therapeutic treatment. Treatment outcomes are assessed with the Outcome Rating Scale (ORS), a four-item self-report instrument measuring client functioning in the area of quality of life. Therapeutic alliance is assessed using the four-item Session Rating Scale (SRS). In FIT the feedback from the client is used to continuous adjustment and improvement of therapy
  Arms: Treatment group

SUMMARY:
Feedback Informed Treatment (FIT) is a systematic feedback method. FIT is based on two simple questionnaires and aims to assess and improve the effectiveness of therapeutic treatment. Treatment outcomes are assessed with the Outcome Rating Scale (ORS), a four-item self-report instrument measuring client functioning in the area of quality of life. Therapeutic alliance is assessed using the four-item Session Rating Scale (SRS). In FIT the feedback from the client is used to continuous adjustment and improvement of therapy. SFI will study the effect of using feedback in social work with floated support in the municipality of Copenhagen. Floating Support is a service that provides housing related support to vulnerable citizens to enable them to maintain their independence in their own home. The project is based on three different types of floating support. The aim of floating support is to improve the citizen's mental, physical and social well-being and thereby makes it more likely that the citizen can live independently at home. The study is a randomized controlled trial in which half of the caseworkers are allocated to be trained in the use of FIT, while the other half serves as a control group and will continue to work as usual. SFI is studying whether FIT can help to improve the impact of the floating support service on the citizen's mental, physical and social well-being and the citizens' likelihood of living in their own homes.

DETAILED DESCRIPTION:
The study was designed as a cluster randomized controlled trial, where the investigators randomized 65 support workers to a treatment group (that used FIT) or a control group (that did not use FIT) at the beginning of the experiment. The investigators used block randomization within each unit to ensure that the number of support workers was evenly distributed between the treatment and control groups within each organizational unit. The investigators generated the random sequence using SAS.

When a support worker resigned during the experiment, another support worker with the same allocation took over the resigned worker's clients. If a new support worker was employed during the experiment in a unit with an even number of workers, the support worker was randomized to either the treatment group or the control group by simple randomization. If the unit had an uneven number of support workers, the new support worker was allocated to a group that ensured the unit kept the same uneven number of treatment and control workers.

The study included clients who had already begun in the support service before the experiment started and clients that started in the support service during the experiment. If a support worker only had one or two contacts with a new client, the client was not included in the study.

The study period was 16 months and ended when FIT was implemented in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Citizens who will receive floating support at the municipality of Copenhagen

Exclusion Criteria:

* Citizens who refuses to get the support. If the caseworkers do not think the citizen will need further support.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1162 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
WHO5 wellbeing scale | 1-15 month after baseline
  The investigators measured the participants wellbeing using the WHO5 wellbeing scale

SECONDARY OUTCOMES:
Drop outs | 1-15 month after baseline
  Number of Drop outs from the floating service
Length of floating support service | 1-15 month after baseline
  The investigators measured treatment duration as the length of the floating support service in the experiment period
Successful support | 1-15 month after baseline
  It floating support service has been successful. Service stopped by caseworker because goal for service reached.
Number of eviction cases | 1-15 month after baseline
  As a measure of possible eviction, the investigators used the mandatory notification sent to the municipality when a citizen living in the public housing sector is subject to an eviction case sent to the Danish bailiff's court.
General health | 1-15 month after baseline
  To measure general health, the investigators used a single global item, that has been used in the SF-36 questionnaire
Social relations | 1-15 month after baseline
  Social relations measured by items from WHO100
Physical wellbeing | 1-15 month after baseline
  Physical wellbeing measured with items from WHO100

CONTACTS AND LOCATIONS:
Overall Officials: Kræn B Jensen, PhD, Study Director — VIVE - The Danish Center for Social Science Research
Locations (1):
- SFI the Danish National Centre for Social Research, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No